CLINICAL TRIAL: NCT00536718
Title: GLACIER: A Study to Investigate the Genetics of LobulAr Carcinoma In Situ in EuRope
Brief Title: Genetics of Women With Lobular Carcinoma in Situ of the Breast
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Research Network (Network)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: NCRN-CRUK-GLACIER; CDR0000566209 (Registry Identifier: PDQ (Physician Data Query)); EU-20760; MREC 06/Q1702/64; CRUK-GLACIER
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer
Keywords: invasive lobular breast carcinoma with predominant in situ component; invasive lobular breast carcinoma; lobular breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Lobular; Breast Carcinoma In Situ | interventions — Gene Expression Profiling; Molecular Diagnostic Techniques; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: molecular diagnostic method
Genetic: polymorphism analysis
Genetic: protein expression analysis
Other: medical chart review
Other: questionnaire administration

SUMMARY:
RATIONALE: Gathering information about genetic changes in patients with lobular carcinoma in situ of the breast may help doctors learn more about the disease and find better methods of treatment.

PURPOSE: This clinical trial is studying the genetics of women with lobular carcinoma in situ of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify inherited variation that predisposes women to develop lobular carcinoma in situ (LCIS) of the breast.
* Identify the frequency of these variants and determine the effect they have on tumor risk.
* Determine how worthwhile it would be to test for these variants in the clinical setting so that those at higher risk could be identified, counseled, and screened.

Secondary

* Analysis of genetic changes within LCIS with the aim of identifying cases of LCIS which may progress to invasive cancer.

OUTLINE: Patients and control participants undergo blood collection. DNA is extracted from blood samples and used to genotype at selected polymorphisms, compare allele frequencies (used to associate alleles with disease) using a genome-wide single nucleotide polymorphism (SNP) screen. Archival tumor samples (if available) from patients are used for DNA-, RNA-, or protein-based analyses.

All participants complete a questionnaire about family history, a brief medical history, and provide epidemiological data to a genetic counselor. Participants identified to be at risk for known hereditary predisposition to cancer will be referred to a clinical genetics service. Individual results of this study are not disclosed to participants.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

PROJECTED ACCRUAL: A total of 2,000 participants (1,000 patients and 1,000 matched controls) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Current or prior diagnosis of lobular carcinoma in situ (LCIS) of the breast, including any of the following cases:

    * Pure LCIS
    * LCIS with subsequent development of invasive breast cancer of any morphological subtype
    * LCIS presenting as an incidental finding together with invasive breast cancer of any morphological subtype
  * Control participant matched for age and ethnicity to each LCIS patient

    * Not affected by LCIS
    * No history of ductal carcinoma in situ of the breast
    * No breast cancer
    * No relative (up to 2nd degree) who has been affected by breast cancer
    * Male or female

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Inherited variation predisposing development of lobular carcinoma in situ (LCIS) of the breast in women
Frequency and effect of variants on tumor risk
Clinical setting variant test value in identifying, counseling and screening those women at higher risk

SECONDARY OUTCOMES:
LCIS genetic changes which may progress to invasive cancer

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Sawyer, MD, Study Chair — London Research Institute; Rebecca Roylance, MD — Barts and the London School of Medicine and Dentistry
Locations (9):
- United Kingdom (9):
  - Basildon University Hospital, Basildon, England
  - Derbyshire Royal Infirmary, Derby, England
  - Leeds General Infirmary, Leeds, England
  - Guy's Hospital, London, England
  - King's College Hospital, London, England
  - London Research Institute, London, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Bronglais District General Hospital, Aberystwyth, Wales
  - Saint Bartholomew's Hospital, London